CLINICAL TRIAL: NCT06942741
Title: A Two-Part Study to Determine Bioequivalence Between the MK-1084 Film-Coated Tablet and Oral-Compressed Tablet and the Effect of Food on the Single-Dose Pharmacokinetics of the MK-1084 Film-Coated Tablet in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Formulation and Food on Calderasib (MK-1084) in Healthy Adult Participants (MK-1084-011)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1084-011; MK-1084-011 (Other: MSD)
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 Calderasib Treatment A (Experimental): Participants will be administered low dose calderasib as an oral-compressed tablet (OCT) on Day 1 under fasted conditions (on an empty stomach after a ≥8-hour fast)
  Interventions: Drug: Calderasib OCT
- Part 1 Calderasib Treatment B (Experimental): Participants will be administered low dose calderasib as a film-coated tablet (FCT) on Day 1 under fasted conditions (on an empty stomach after a ≥8-hour fast)
  Interventions: Drug: Calderasib FCT
- Part 2 Calderasib Treatment C (Experimental): Participants will be administered higher dose calderasib as a FCT on Day 1 under fasted conditions (on an empty stomach after a ≥8-hour fast)
  Interventions: Drug: Calderasib FCT
- Part 2 Calderasib Treatment D (Experimental): Participants will be administered higher dose calderasib as a FCT on Day 1 under fed conditions (after a high-fat meal)
  Interventions: Drug: Calderasib FCT

INTERVENTIONS:
Drug: Calderasib OCT — Oral tablet
  Other Names: MK-1084 OCT
  Arms: Part 1 Calderasib Treatment A
Drug: Calderasib FCT — Oral tablet
  Other Names: MK-1084 FCT
  Arms: Part 1 Calderasib Treatment B; Part 2 Calderasib Treatment C; Part 2 Calderasib Treatment D

SUMMARY:
This study has 2 parts. Researchers want to learn what happens to calderasib in a healthy person's body over time in both parts. The goals of the study are:

* In Part 1, to compare what happens to calderasib in a person's blood when it is taken as 2 different types of oral tablets
* In Part 2, to learn what happens to calderasib in a person's blood when it is taken on an empty stomach or after a meal

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

- Has a body mass index ≥18.0 and ≤32.0 kg/m^2

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has a history or presence of a clinically significant medical or psychiatric condition or disease
* Has a history of cancer (malignancy)
* Has positive results for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-06-22 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Parts 1 and 2: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-last) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the AUC0-last of calderasib.
Parts 1 and 2: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUC0-inf) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the AUC0-inf of calderasib.
Parts 1 and 2: Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24) of Calderasib | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the AUC0-24 of calderasib.
Parts 1 and 2: Maximum Plasma Concentration (Cmax) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the Cmax of calderasib.
Parts 1 and 2: Plasma Concentration of Calderasib at 24 Hours Postdose (C24) | At designated timepoints (up to 24 hours postdose)
  Blood samples will be collected to determine the C24 of calderasib.
Parts 1 and 2: Time to Maximum Plasma Concentration (Tmax) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the Tmax of calderasib.
Parts 1 and 2: Apparent Terminal Half-life (t1/2) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the t1/2 of calderasib.
Parts 1 and 2: Apparent Clearance (CL/F) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the CL/F of calderasib.
Parts 1 and 2: Apparent Volume of Distribution During Terminal Phase (Vz/F) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the Vz/F of calderasib.
Part 2: Plasma Lag Time (tlag) of Calderasib | At designated timepoints (up to approximately 2 days postdose)
  Blood samples will be collected to determine the tlag of calderasib.

SECONDARY OUTCOMES:
Parts 1 and 2: Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 7 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be reported
Parts 1 and 2: Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 1 week
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue from the study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion ( Site 0001), Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/